CLINICAL TRIAL: NCT06592248
Title: Evaluation of a New Bi-Condylar Total Knee Prosthesis (TKP) With All-Ceramic Friction
Brief Title: Evaluation of a New Bi-Condylar Total Knee Prosthesis (TKP) With All-Ceramic Friction (The Forgotten Knee)
Acronym: ForgottenKne
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190284; 2020-A02892-37 (Other: IDRCB)
Record Dates: First submitted 2024-07-16; First posted 2024-09-19 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Prosthesis; Ceramic on ceramic bearing
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: * Validation of the concept
  * Absence of added risks after implementation
  * Measurement of fibrous tissue formed by MRI examination
  Inclusion will be done by sequencing in 2 steps:
  * Inclusion of 2 patients with implementation of the experimental MD with a post-operative follow-up of 3 months,
  * if no SAE linked to the experimental MD is detected, the inclusions will continue until the 5th patient with experimental DM,
  * In the event of notification of an SAE linked to the experimental MD according to the investigator in the first 2 patients, within the first 3 months, the research will be stopped prematurely
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CocKnee (Experimental): Implementation of CocKnee
  Interventions: Device: Coc Knee

INTERVENTIONS:
Device: Coc Knee — Implementation of a ceramic on ceramic knee prosthesis

SUMMARY:
The results of TKP (Total Knee Prosthesis) are satisfactory but do not reach those of THP (Total Hip Prosthesis) in terms of indolence and function. By using an all-ceramic friction torque, identical to that of the hip, the promotor of this Clinical Investigation expects to obtain an improvement in term of indolence, ability to perform heavy activities, knee stability and an improvement in the long-term survival of TKP, while at the same time, a decrease in the rate of re-intervention in young patients.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the all-ceramic knee prosthesis, according to clinical and radiological criteria of usual follow-up of a TKP for knee osteoarthritis, at 12 months.

Evaluation of clinical and radiographic endpoints at 12 months:

- Clinical: functional scores (Oxford and International Knee Society IKS), pain (from 0 to 6, better to worse outcome), knee mobility in flexion and extension (degrees), frontal and sagittal stability (in degrees and mm), joint sounds, Forgotten Joint Score (FJS).

The scores are mostly qualitative and all of them will be globally evaluated by the investigator regarding to the patient status.

-Radiographic: X-rays of the front and profile of the prosthesis, positioning of the implants (angle, axis), existence of borders (bone cement, prosthesis cement), presence of osteolysis or any notable element.

MRI will be performed to evaluate the creation of a specific fibrous tissue around the joint that is expected with a ceramic on ceramic bearing.

ELIGIBILITY:
Inclusion Criteria:

* Previously active adult under 70 years of age with disabling knee osteoarthritis resistant to medical treatments (anti-inflammatories, infiltrations, analgesics), with a frontal deformity < 10° for a primary implantation
* Written informed consent by the patient
* Patients affiliated to the French social security system

Exclusion Criteria:

* Knee deformity > 10
* Obesity (BMI > 30)
* Inflammatory rheumatism
* History of infection
* Poor skin coverage at the knee joint
* Known allergy to the materials used and/or anesthetic used in the surgery
* Repeated falls, major neurological disorders, mental or neuromuscular disorders which can be a source of post-operative complications
* Significant functional deficit of the collateral ligaments
* Positive serum or urine pregnancy test for woman with child bearing potential. Pregnancy or within 48 hours post-partum or breast feeding women
* Phobic patient refusing to have an MRI
* Patient with a contraindication to have an MRI (active medical devices, metal implants, etc.)
* Patient under legal protection
* Patient participating in another Clinical Investigation
* Post fracture osteoarthritis
* Osteoporosis
* Anatomical configuration not allowing the implant to be fixed (depending on size constraints)
* Disabling comorbidity upon any resumption of physical activity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical endpoint 1(Oxford score) at 12 months | 1 year
  Clinical 1 :
  Oxford functional score : 12 (good) to 60 (bad) 12 questions (1 normal to 5 discomfort )
Evaluation of clinical endpoint 2 (IKS score) at 12 months | 1 year
  Clinical 2 :
  International Knee Society (IKS) score :
  * objective component (symptoms) 25 points
  * subjective component:
    * expectation (pre or post surgery) 15 points
    * satisfaction 40 points
    * function 100 points
Evaluation of clinical endpoint 3 (Forgotten Joint score) at 12 months | 1 year
  Clinical 3 :
  Forgotten Joint Score (FJS) :
  12 questions (0 normal to 4 discomfort ) = Total then FJScore = 100 - (Total x 25)
Evaluation of clinical endpoint 4 (Joint sounds) at 12 months | 1 year
  Clinical 4:
  Joint sounds :
  5 questions, no score
Evaluation of clinical endpoint 5 (Pain) at 12 months | 1 year
  Clinical 5:
  Pain : 0 to 6
Evaluation of clinical endpoint 6 (Knee mobility) at 12 months | 1 year
  Clinical 6:
  Knee mobility :
  Flexion (°) Extension (°)
Evaluation of clinical endpoint 7 (Knee stability) at 12 months | 1 year
  Clinical 7:
  Knee stability :
  Frontal (° and mm) Sagittal (° and mm)
Evaluation of radiographic endpoints at 12 months | 1 year
  Radiographic :
  X-rays of the front and profile of the prosthesis : positioning of the implants (angle, axis), existence of borders (bone cement, prosthesis cement), presence of osteolysis or any notable element.

SECONDARY OUTCOMES:
Evaluation of clinical endpoint 1 (Oxford score) at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Clinical 1 :
  Oxford functional score : 12 (good) to 60 (bad) 12 questions (1 normal to 5 discomfort )
Evaluation of clinical endpoint 2 (IKS score) at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Clinical 2 :
  International Knee Society (IKS) score :
  * objective component (symptoms) 25 points
  * subjective component:
    * expectation (pre or post surgery) 15 points
    * satisfaction 40 points
    * function 100 points
Evaluation of clinical endpoint 3 (FJ Score) at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Clinical 3 :
  Forgotten Joint Score (FJS) :
  12 questions (0 normal to 4 discomfort ) = Total then FJScore = 100 - (Total x 25)
Evaluation of clinical endpoint 4 (Joint sounds) at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Clinical 4 :
  Joint sounds :
  5 questions, no score
Evaluation of clinical endpoint 5 (Pain) at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Clinical 5 :
  Pain : 0 to 6
Evaluation of clinical endpoint 6 (Knee mobility) at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Clinical 6 :
  Knee mobility :
  Flexion (°) Extension (°)
Evaluation of clinical endpoint 7 (Knee stability) at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Clinical 7 :
  Knee stability :
  Frontal (° and mm) Sagittal (° and mm)
Evaluation of radiographic endpoints at 3 and 6 months and physical capabilities of the patient | 3 and 6 months
  Radiographic :
  X-rays of the front and profile of the prosthesis : positioning of the implants (angle, axis), existence of borders (bone cement, prosthesis cement), presence of osteolysis or any notable element.
Evaluation of fibrous tissue | 1 year
  Evaluation of fibrous tissue around the prosthesis:
  Performance of ultrasounds and MRI at 3, 6 and 12 months postoperatively, allowing to evaluate and measure (in mm) the thickness and progression of fibrous tissue around the prosthesis.
Validation of the ancillary equipment used and the prosthesis surgical technique | 1 year
  Notification of any malfunction noticed during the use of ancillary equipment

CONTACTS AND LOCATIONS:
Overall Officials: Pascal BIZOT, MD, Pr, Principal Investigator — APHP; Laurent SEDEL, MD, Pr, Study Director — CC/ Contact
Locations (1):
- Hôpital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: No